CLINICAL TRIAL: NCT03915730
Title: The Effect of Smoking on Gingival Crevicular Fluid Peptidoglycan Recognition Protein-1 Level Following Initial Periodontal Therapy in Chronic Periodontitis
Brief Title: Smoking and Peptidoglycan Recognition Protein-1 and Initial Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Meltem Karsiyaka Hendek, Assistant Professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/026
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Smoking, Cigarette
Keywords: Chronic periodontitis; gingival crevicular fluid; initial periodontal therapy; peptidoglycan recognition proteins; smoking
MeSH Terms: conditions — Cigarette Smoking; Chronic Periodontitis; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Smokers with chronic periodontitis (Experimental): Patients who had teeth with 30% periodontal bone loss, presence of at least two nonadjacent sites per quadrant with probing pocket depths of ≥5 mm, and bleeding on probing were assigned as chronic periodontitis group Patients who have smoked for at least 10 years and a minimum of 10 cigarettes per day were assigned as current smokers.
  Interventions: Other: Initial periodontal therapy
- Non-smokers with chronic periodontitis (Experimental): Patients who had teeth with 30% periodontal bone loss, presence of at least two nonadjacent sites per quadrant with probing pocket depths of ≥5 mm, and bleeding on probing were assigned as chronic periodontitis group Never smoked patients were included into the nonsmoker group
  Interventions: Other: Initial periodontal therapy
- Smokers with periodontal healthy (No Intervention): Individuals were diagnosed periodontally healthy as without attachment loss, periodontal disease history, whole mouth bleeding scores of <10% and a probing depth of ≤3 mm Patients who have smoked for at least 10 years and a minimum of 10 cigarettes per day were assigned as current smokers.
- Non-smokers with periodontal healthy (No Intervention): Individuals were diagnosed periodontally healthy as without attachment loss, periodontal disease history, whole mouth bleeding scores of <10% and a probing depth of ≤3 mm Never smoked patients were included into the nonsmoker group

INTERVENTIONS:
Other: Initial periodontal therapy — Scaling and root planing and polishing with specific curettes were performed to patients with CP and oral hygiene education was provided to each patient.
  Arms: Non-smokers with chronic periodontitis; Smokers with chronic periodontitis

SUMMARY:
A total of 40 patients with CP (20 smokers (S+CP) and 20 nonsmokers (S-CP)) and 40 periodontally healthy subjects (20 smokers (S+PH) and 20 nonsmokers (S-PH)), comprising 80 subjects, were included in this study. Baseline GCF samples were obtained from all subjects and clinical periodontal measurements, including probing depth (PD), clinical attachment level (CAL), plaque index (PI), and gingival index (GI), were recorded. In patients who had received initial periodontal therapy, GCF samples were obtained and all clinical periodontal measurements were recorded again during the 6th-8th weeks. GCF PGRP-1 levels were analyzed by enzyme-linked immunosorbent assay.

DETAILED DESCRIPTION:
Peptidoglycan recognition proteins (PGRPs) are one of the antimicrobial peptides that play a role in innate immunity and act against the bacterial cell wall. Smoking is the most important environmental risk factor for periodontitis. This study determined the effect of smoking on PGRP-1 levels in gingival crevicular fluid (GCF) in smokers and nonsmokers with chronic periodontitis (CP) following initial periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe chronic periodontitis
* Clinical diagnosis of periodontal health

Exclusion Criteria:

* have any systemic disease,
* to be alcohol consumer,
* to receive any periodontal therapy in the past 6 months,
* to take any drugs regularly
* to be pregnant and/or lactate.

Ages: 22 Years to 56 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in peptidoglycan recognition protein-1 | Baseline and 3 months
  Total amount of Peptidoglycan Recognition Protein-1 (µg) in gingival crevicular fluid

SECONDARY OUTCOMES:
Change in periodontal clinical parameter | Baseline and 3 months
  Clinical attachment level (mm) (from cemento-enamel junction to the base of periodontal pocket)